CLINICAL TRIAL: NCT04292223
Title: A 16-Week Open-Label Study of the Effects of Treatment With Pimavanserin on Activities of Daily Living in Subjects With Parkinson's Disease Psychosis
Brief Title: Open-Label Study With Pimavanserin on Activities of Daily Living in Subjects With Parkinson's Disease Psychosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACP-103-063
Record Dates: First submitted 2020-02-28; First posted 2020-03-03 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-12

CONDITIONS: Parkinson Disease Psychosis
MeSH Terms: interventions — pimavanserin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Drug - Pimavanserin (Experimental): Pimavanserin 34 mg administered orally
  Interventions: Drug: Pimavanserin

INTERVENTIONS:
Drug: Pimavanserin — Pimavanserin 34 mg (provided as 1×34 mg capsule), administered orally, once daily for 16 weeks
  Other Names: NUPLAZID

SUMMARY:
To assess the effect of pimavanserin on the activities of daily living in subjects with Parkinson's Disease Psychosis

DETAILED DESCRIPTION:
This study will be conducted as a 16-week, multi-center, single-arm, open-label study. Pimavanserin will be administered at a dose of 34 mg to approximately 50 subjects with PDP

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects at least 40 years of age
2. Has a Mini-Mental State Examination (MMSE) score ≥19 at Screening
3. Has a diagnosis of idiopathic Parkinson's disease (PD)
4. Has psychotic symptoms that may impair function and are severe enough to warrant treatment with an antipsychotic agent
5. Psychotic symptoms developed after the onset of symptoms of PD
6. If the subject is female, she must not be pregnant or breastfeeding. She must also be of non-childbearing potential (defined as either surgically sterilized or at least 1 year postmenopausal) OR must agree to use TWO clinically acceptable methods of contraception.

Exclusion Criteria:

1. Has atypical parkinsonism (Parkinson's plus, multiple system atrophy [MSA], progressive supranuclear palsy [PSP]), or secondary parkinsonism variants such as tardive or medication induced parkinsonism
2. Has undergone ablative procedures such as a pallidotomy, thalamotomy, or treatment with focused ultrasound, or has an implanted deep brain stimulator
3. Has current evidence of an unstable neurological, cardiovascular, respiratory, gastrointestinal, renal, hepatic, hematologic, or other medical or psychiatric disorder, including cancer or malignancies that, in the judgment of the Investigator, would jeopardize the safe participation of the subject in the study or significantly interfere with the conduct or interpretation of the study
4. Has a history of myocardial infarction, unstable angina, acute coronary syndrome, or cerebrovascular accident within the last 6 months prior to Screening
5. Has any of the following:

   1. greater than New York Heart Association (NYHA) Class 2 congestive heart failure
   2. Grade 2 or greater angina pectoris (by Canadian Cardiovascular Society Angina Grading Scale)
   3. sustained ventricular tachycardia
   4. ventricular fibrillation
   5. torsades de pointes
   6. syncope due to an arrhythmia
   7. an implantable cardiac defibrillator
6. Has a known personal or family history of long QT syndrome or family history of sudden cardiac death
7. Requires treatment with a medication or other substance that is prohibited by the protocol
8. Has a body mass index (BMI) <18.5 kg/m2 or >35 kg/m2 at Screening or Baseline or known unintentional clinically significant weight loss (i.e., ≥7%) over past 6 months
9. Is suicidal at Screening or Baseline
10. Has a history of a significant psychotic disorder prior to or concomitantly with the onset of PD including, but not limited to, schizophrenia or bipolar disorder
11. Had dementia prior to or concomitantly with the onset of motor symptoms of PD
12. Positive COVID-19 polymerase chain reaction (PCR) or antigen result in the last 2 weeks prior to screening
13. Is judged by the Investigator or the Medical Monitor to be inappropriate for the study for any reason

Additional inclusion/exclusion criteria apply. Subjects will be evaluated at screening to ensure that all criteria for study participation are met.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2022-04-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Movement Disorders Center of Arizona, Scottsdale, Arizona
  - Neurology Center of North Orange County, Fullerton, California
  - Premier Clinical Research Institute, Inc., Miami, Florida
  - Global Health Research Center, Inc., Miami Lakes, Florida
  - Quantum Laboratories, Inc., Pompano Beach, Florida
  - Parkinson's Disease Treatment Center of Southwest Florida, Port Charlotte, Florida
  - Accel Research Sites - Brain and Spine Institute, Port Orange, Florida
  - Infinity Clinical Research, LLC, Sunrise, Florida
  - Premiere Research Institute at Palm Beach Neurology, West Palm Beach, Florida
  - AU Movement and Memory Disorders, Augusta, Georgia
  - Maine Medical Partners Neurology, Scarborough, Maine
  - Wentworth Health Partners Coastal Neurology Services, Dover, New Hampshire
  - Bio Behavioral Health, Toms River, New Jersey
  - Neurology Diagnostics, Inc., Dayton, Ohio
  - The Orthopedic Foundation, New Albany, Ohio
  - Central States Research, Tulsa, Oklahoma
  - KCA Neurology, Franklin, Tennessee
  - Neurological Associates of North Texas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Evidente VGH, DeKarske D, Coate B, Abler V. The effects of treatment with pimavanserin on activities of daily living in patients with Parkinson's disease psychosis: a 16-week, single-arm, open-label study. Ther Adv Neurol Disord. 2024 Mar 11;17:17562864241228350. doi: 10.1177/17562864241228350. eCollection 2024. PMID 38476466

RESULTS

PARTICIPANT FLOW:
Groups:
- Pimavanserin 34 mg: Pimavanserin 34 mg (one capsule of 34 mg dose strength) taken orally once daily
Period: Overall Study
Arm/Group | Pimavanserin 34 mg
Started | 29
Completed | 24
Not Completed | 5
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1
Not completed — Noncompliance with study drug | 2
Not completed — Patient moved out of the state | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pimavanserin 34 mg
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.2 (8.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 28
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 16 in Modified Functional Status Questionnaire (mFSQ) Total Score
Description: The mFSQ is a self-administered questionnaire. It comprises 34 core items that produce 6 summary scale scores (i.e. basic activities of daily living (ADL); intermediate ADL; psychological function and mental health; work performance, social activity, and quality of interaction) and 6 single-item scores (work situation; days/month in bed due to illness/injury; days/month when illness/injury reduced activities normally performed for half a day; satisfaction with sexual relationship; satisfaction with health; frequency of social interaction).
  The mFSQ is calculated as the unweighted mean of predefined subscale scores. The maximum mFSQ total score is 100, with higher scores indicating better functional status. The minimum score is 0 and the maximum score is 100.
Time Frame: 16 weeks
Population: All patients enrolled and with baseline mFSQ value
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin 34 mg
Number analyzed (Participants) | 28
score on a scale | 14.0 (2.50)
Statistical Analysis 1: Comparison: Pimavanserin 34 mg; Test type: Other — Comparison of the 16-week value with the baseline value; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 14.0, 95% CI 2-sided [8.8 to 19.3], Standard Error of Mean 2.50

2. Secondary Outcome: Change From Baseline to Week 16 on the Schwab and England Activity of Daily Living (ADL) Scale, Caregiver and Patient Versions
Description: The Schwab & England ADL Scale is a scale ranging from 0% to 100% scale with 10% intervals, where 100% is "Completely independent. Unaware of difficulty" and 0% is "Vegetative functions such as swallowing, bladder and bowel functions are not functioning. Bedridden"
Time Frame: 16 Weeks
Population: All patients enrolled and with baseline mFSQ value
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin 34 mg
Number analyzed (Participants) | 28
score on a scale
  Patient version | 3.4 (2.97)
  Caregiver version | 2.6 (2.75)

3. Secondary Outcome: Change From Baseline to Week 16 on the Movement Disorders Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Parts I and II
Description: The MDS-UPDRS is a battery of motor and behavioral indices. MDS-UPDRS Part I assesses non-motor aspects of experiences of daily living (EDL) and consists of 13 items (6 investigator assessed; 7 patient assessed, each scored on a 5-point Likert scale). The total score is the sum of the 13 individual items. The highest score is 52, higher scores mean more severe impact of the disease on non-motor aspects of ADL and the lowest score is 0. In Part 1, a lower score is better while a higher score is worse.
  Part II assesses motor aspects of EDL and consists of 13 items (all patient assessed, each on a 5-point Likert scale). The highest score is 52, higher scores mean more severe impact of the disease on motor aspects of ADL and the lowest score is 0. In Part 2, a lower score is better while a higher score is worse.
Time Frame: 16 Weeks
Population: All patients enrolled and with baseline mFSQ value
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin 34 mg
Number analyzed (Participants) | 28
score on a scale
  MDS-UPDRS Part I | -0.63 (0.97)
  MDS-UPDRS Part II | -2.6 (0.98)

4. Secondary Outcome: Week 16 Clinical Global Impression - Improvement (CGI-I) Score for Hallucinations and Delusions
Description: The CGI-I is a clinician-rated, 7-point scale to rate the improvement in patient symptoms at the time of assessment, relative to the symptoms at baseline. Severity ratings are based on the behavioral domains of hallucinations and delusions. The score ranges from 1=very much improved to 7=very much worse. Higher scores denote more severe symptoms of hallucinations and delusions
Time Frame: 16 Weeks
Population: All patients enrolled and with baseline mFSQ value
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin 34 mg
Number analyzed (Participants) | 28
score on a scale | 1.9 (0.17)

5. Secondary Outcome: Change From Baseline to Week 16 on the Clinical Global Impression - Severity of Illness (CGI-S) Score for Hallucinations and Delusions
Description: The CGI-S scale is a clinician-rated, 7-point scale to rate the severity of patient neuropsychiatric symptoms at the time of assessment using the Investigator's judgment and past experience with patients who have the same disorder. Severity ratings aree based on the behavioral domains of hallucinations and delusions.The score ranges from 1=normal, not at all ill to 7=among the most extremely ill patients. Higher scores denote more severe symptoms of hallucinations and delusions.
Time Frame: 16 Weeks
Population: All patients enrolled and with baseline mFSQ value
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin 34 mg
Number analyzed (Participants) | 28
score on a scale | -1.5 (0.25)

6. Secondary Outcome: Patient Global Impression of Improvement (PGI-I) Score for Hallucinations and Delusions at Week 16
Description: The PGI-I is a global index to rate the response of a condition to a therapy. Patients have to rate their current symptoms, compared with baseline. Responses range from 1=very much better to 7=very much worse. Severity ratings are based on the behavioral domains of hallucinations and delusions.
Time Frame: 16 Weeks
Population: All patients enrolled and with baseline mFSQ value
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin 34 mg
Number analyzed (Participants) | 28
score on a scale | 2.0 (0.22)

ADVERSE EVENTS:
Time Frame: From informed consent through the Safety Follow-up period, for a total of up to 181 day (i.e. Screening period of 3 to 35 days; Open-label Treatment period of 16 weeks; and Safety Follow-up period of 30 to 34 days)
Arm/Group | Pimavanserin 34 mg
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 3/29
Other Adverse Events (participants affected / at risk) | 9/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pimavanserin 34 mg (N=29)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pimavanserin 34 mg (N=29)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Inflammation (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Peripheral swelling (General disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Cellulitis (Infections and infestations) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3)
Sinus headache (Nervous system disorders) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator may publish the study results, relative to his/her own patients, only after review, comment and approval by the sponsor. No publication of confidential information shall be made without the sponsor's prior written consent. At least 60 days prior to submitting a manuscript or prior to any public presentation, a copy of the manuscript or presentation will be provided to the sponsor for review and comment. The sponsor has 60 days to review and comment.

DOCUMENTS (2):
  • Study Protocol (2021-05-20): https://cdn.clinicaltrials.gov/large-docs/23/NCT04292223/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-28): https://cdn.clinicaltrials.gov/large-docs/23/NCT04292223/SAP_001.pdf